CLINICAL TRIAL: NCT03073005
Title: Use of Simulation to Improve Ventricular Assist Device Self-management
Brief Title: Use of Simulation to Improve VAD Self-management
Acronym: SimVAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Jeffrey Barsuk, Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STU00203530; 5R21NR016745-02 (NIH)
Record Dates: First submitted 2017-02-20; First posted 2017-03-08 (Actual); Results first posted 2021-05-10 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Heart Failure
Keywords: ventricular assist device (VAD); heart failure; simulation
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional VAD training (No Intervention): Patients and caregivers will receive traditional training for their VAD via a video produced by the VAD manufacturer.
- Simulation-based VAD training (Experimental): Patients and caregivers will receive traditional training for their VAD via a video produced by the VAD manufacturer and then participate in simulation-based mastery learning for VAD management
  Interventions: Other: Simulation-based Mastery Learning (SBML)

INTERVENTIONS:
Other: Simulation-based Mastery Learning (SBML) — The SBML training group will first 1) watch the VAD video, then 2) participate in a SBML intervention using the simulator for a) driveline exit site sterile dressing changes; b) performing controller self-tests; c) changing power sources; d) troubleshooting emergent VAD-related malfunction; and e) recognizing specific signs and symptoms requiring immediate contact with the VAD team.
  Arms: Simulation-based VAD training

SUMMARY:
This study will evaluate the performance of a curriculum using medical simulators to train patients with advanced heart failure and their caregivers to master the self-management of ventricular assist devices (a device implanted into the heart to help circulate the blood). The investigators expect this training will improve self-management skills, and reduce VAD-related infections and re-hospitalizations. In addition to providing innovative training to the patients and their caregivers, the study will advance our knowledge of the effects of simulation-based training on patient self-management and safety.

ELIGIBILITY:
Patient Inclusion Criteria:

* being a previous or current VAD implantation patient,
* age >18,
* English-speaking,
* receiving implantation and VAD care at Northwestern Memorial Hospital (NMH),
* meet hospital criteria for VAD implantation.

Caregiver inclusion criteria:

* being a caregiver identified by a previous or current VAD implantation patient,
* age >18, and
* English-speaking.

Exclusion Criteria:

* Vulnerable populations of patients will not be included in this study (including fetuses, neonates, children, pregnant women, prisoners, mentally retarded or incompetent individuals, institutionalized individuals, or individuals unable to give consent due to their medical condition). Fetuses and neonates are not the focus of our study.
* Pregnant women will not be included since pregnancy is a contraindication to VAD implantation It is possible that VAD caregivers may be pregnant at the time of the study.
* Patients with mental retardation, mental incompetence, or patients who are unable to give consent due to their medical condition will not be included as they will not be able to complete measures.
* Lastly, institutionalized individuals will not be included as access will be a problem, and these individuals are rarely referred for VAD implantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Barsuk, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Barsuk JH, Wilcox JE, Cohen ER, Harap RS, Shanklin KB, Grady KL, Kim JS, Nonog GP, Schulze LE, Jirak AM, Wayne DB, Cameron KA. Simulation-Based Mastery Learning Improves Patient and Caregiver Ventricular Assist Device Self-Care Skills: A Randomized Pilot Trial. Circ Cardiovasc Qual Outcomes. 2019 Oct;12(10):e005794. doi: 10.1161/CIRCOUTCOMES.119.005794. Epub 2019 Oct 11. PMID 31601111

RESULTS

PARTICIPANT FLOW:
Groups:
- Traditional VAD Training (Patients): Patients will receive traditional training for their VAD via a video produced by the VAD manufacturer.
- Traditional VAD Training (Caregivers): Caregivers will receive traditional training for their VAD via a video produced by the VAD manufacturer.
- Simulation-based VAD Training (Patients): Patients will receive traditional training for their VAD via a video produced by the VAD manufacturer and then participate in simulation-based mastery learning for VAD management
  Simulation-based Mastery Learning (SBML): The SBML training group will first 1) watch the VAD video, then 2) participate in a SBML intervention using the simulator for a) driveline exit site sterile dressing changes; b) performing controller self-tests; c) changing power sources; d) troubleshooting emergent VAD-related malfunction; and e) recognizing specific signs and symptoms requiring immediate contact with the VAD team.
- Simulation-based VAD Training (Caregivers): Caregivers will receive traditional training for their VAD via a video produced by the VAD manufacturer and then participate in simulation-based mastery learning for VAD management
  Simulation-based Mastery Learning (SBML): The SBML training group will first 1) watch the VAD video, then 2) participate in a SBML intervention using the simulator for a) driveline exit site sterile dressing changes; b) performing controller self-tests; c) changing power sources; d) troubleshooting emergent VAD-related malfunction; and e) recognizing specific signs and symptoms requiring immediate contact with the VAD team.
Period: Overall Study
Arm/Group | Traditional VAD Training (Patients) | Traditional VAD Training (Caregivers) | Simulation-based VAD Training (Patients) | Simulation-based VAD Training (Caregivers)
Started | 33 | 37 | 36 | 37
Received Initial Training | 29 (29 pairs (29 patients plus their caregivers)) | 29 | 33 (33 pairs (33 patients plus their caregivers)) | 33
Completed (Completed entire protocol thru discharge testing) | 25 (25 pairs (25 patients plus their caregivers)) | 25 | 24 (24 pairs (24 patients plus their caregivers)) | 24
Not Completed | 8 | 12 | 12 | 13
Not completed — Death | 6 | 0 | 7 | 0
Not completed — caregiver withdrew bc of pt death | 0 | 6 | 0 | 7
Not completed — Lost to Follow-up | 2 | 2 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 4 | 4 | 4

BASELINE CHARACTERISTICS:
Population: in order to be considered for final analysis both the patient participant plus their caregiver (pairs) must still be enrolled in the study
Groups:
- Traditional VAD Training (Patients); Traditional VAD Training (Caregivers): Patients and caregivers will receive traditional training for their VAD via a video produced by the VAD manufacturer.
- Simulation-based VAD Training (Patients); Simulation-based VAD Training (Caregivers): Patients and caregivers will receive traditional training for their VAD via a video produced by the VAD manufacturer and then participate in simulation-based mastery learning for VAD management
  Simulation-based Mastery Learning (SBML): The SBML training group will first 1) watch the VAD video, then 2) participate in a SBML intervention using the simulator for a) driveline exit site sterile dressing changes; b) performing controller self-tests; c) changing power sources; d) troubleshooting emergent VAD-related malfunction; and e) recognizing specific signs and symptoms requiring immediate contact with the VAD team.
- Total: Total of all reporting groups
Arm/Group | Traditional VAD Training (Patients) | Traditional VAD Training (Caregivers) | Simulation-based VAD Training (Patients) | Simulation-based VAD Training (Caregivers) | Total
Number analyzed (Participants) | 33 | 37 | 36 | 37 | 143
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.91 (13.25) | 53.43 (14.95) | 51.33 (14.54) | 55.28 (12.68) | 53.71 (13.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 30 | 10 | 27 | 76
  Male | 24 | 7 | 26 | 10 | 67
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 6 | 4 | 15
  Not Hispanic or Latino | 30 | 35 | 30 | 33 | 128
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1 | 2
  Asian | 1 | 1 | 2 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 11 | 14 | 12 | 12 | 49
  White | 19 | 21 | 20 | 22 | 82
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 1 | 1 | 5
Region of Enrollment [Number; unit: participants]
  United States | 33 | 37 | 36 | 37 | 143
Baseline VAD Checklist Skills [Median (Inter-Quartile Range); unit: percent of items correct on checklist] — Baseline skills assessed via checklists for SBML-trained patients and caregivers ONLY on controller change, power source change and dressing change (caregiver only). Scored in terms of percent checklist items correct. Population: ONLY SBML-trained patients and caregivers took a baseline exam. Traditionally-trained patients and caregivers scores in the study were considered their "baseline". Those are reported in the outcomes section.
  *dressing change is for caregivers only
  percent of items correct on checklist
    Controller change: number analyzed (Participants) | 0 | 0 | 36 | 37 | 73
    Controller change |  |  | 21.42 [1.79 to 33.93] | 28.57 [21.43 to 66.07] | 24.04 [9.82 to 48.21]
    Power source change: number analyzed (Participants) | 0 | 0 | 36 | 37 | 73
    Power source change |  |  | 22.22 [0 to 66.67] | 76.39 [38.46 to 88.89] | 55.56 [0 to 88.89]
    Dressing change: number analyzed (Participants) | 0 | 0 | 0 | 37 | 37
    Dressing change |  |  |  | 23.44 [10.16 to 32.01] | 23.44 [10.16 to 32.01]

OUTCOME MEASURES:

1. Primary Outcome: Comparisons of VAD-care Checklist Assessment on the Patient and Written Examination Scores Between SBML and Usual Training Groups
Description: The investigators will compare the performance of the SBML intervention group to the usual VAD training group during actual VAD care activities (controller change, power source change and dressing change) plus a written examination. Only caregivers were assessed on dressing change as patients do not independently complete this task.
Time Frame: 3 months
Population: Patient and caregiver pairs were included if both the patient and their caregiver completed training and assessments through discharge testing. (*Note- Only caregivers were assessed on dressing change as patients do not independently complete this task.)
Measure: Median (Inter-Quartile Range); unit: percentage of checklist items correct
Arm/Group | Traditional VAD Training (Patients) | Traditional VAD Training (Caregivers) | Simulation-based VAD Training (Patients) | Simulation-based VAD Training (Caregivers)
Number analyzed (Participants) | 25 | 25 | 24 | 24
percentage of checklist items correct
  Written examination | 100 [97.1 to 100] | 97.1 [97.1 to 100] | 100 [97.1 to 100] | 100 [97.1 to 100]
  Controller change | 92.9 [78.6 to 100] | 100 [100 to 100] | 100 [100 to 100] | 100 [100 to 100]
  Power source change | 88.9 [88.9 to 88.9] | 88.9 [88.9 to 96.2] | 100 [100 to 100] | 100 [100 to 100]
  Dressing change: number analyzed (Participants) | 0 | 25 | 0 | 24
  Dressing change |  | 81.3 [68.8 to 87.5] |  | 100 [100 to 100]

2. Secondary Outcome: Infections and Re-hospitalizations up to 3 Months After VAD Implant
Description: All VAD related driveline infections and re-hospitalizations between the SBML intervention group as compared to the usual VAD training group
Time Frame: 3 months after discharge
Population: This outcome is for patients only
Measure: Count of Participants; unit: Participants
Arm/Group | Traditional VAD Training (Patients) | Simulation-based VAD Training (Patients)
Number analyzed (Participants) | 25 | 24
Participants
  Infections | 6 | 0
  Re-hospitalizations | 20 | 15

3. Secondary Outcome: Self-management Skill Decay in the Five Domains
Description: The investigators will measure the change in skill decay on the patient from 0 (time of implant), one and three months using VAD self-management checklists (controller change, power source change and dressing change) throughout the study period.
Time Frame: 1 month and 3 months after discharge (*1 month SBML-trained only)
Population: Of the 49 patient and caregiver pairs who completed discharge testing, 15 patient and caregiver pairs in the SBML group completed 1 month and 3 month followup testing and 20 pairs in the usual care group completed 3 month follow-up testing only.
Measure: Median (Inter-Quartile Range); unit: percentage of checklist items correct
Arm/Group | Traditional VAD Training (Patients) | Traditional VAD Training (Caregivers) | Simulation-based VAD Training (Patients) | Simulation-based VAD Training (Caregivers)
Number analyzed (Participants) | 20 | 20 | 15 | 15
percentage of checklist items correct
  One month controller change: number analyzed (Participants) | 0 | 0 | 15 | 15
  One month controller change |  |  | 100 [78.57 to 100] | 100 [100 to 100]
  One month power source change: number analyzed (Participants) | 0 | 0 | 15 | 15
  One month power source change |  |  | 100 [100 to 100] | 100 [100 to 100]
  One month dressing change: number analyzed (Participants) | 0 | 0 | 0 | 15
  One month dressing change |  |  |  | 100 [90.63 to 100]
  3 month controller change | 85.71 [62.50 to 100] | 78.57 [28.57 to 100] | 100 [78.57 to 100] | 100 [100 to 100]
  3 month power source change | 88.89 [88.89 to 97.22] | 88.89 [88.89 to 88.89] | 100 [100 to 100] | 100 [100 to 100]
  3 month dressing change: number analyzed (Participants) | 0 | 20 | 0 | 15
  3 month dressing change |  | 78.13 [67.99 to 86.42] |  | 100 [93.75 to 100]

4. Secondary Outcome: Comparisons of Self-confidence Between Groups
Description: Simulation-based Mastery Learning (SBML) Trained and Usual Trained Patient and Caregiver Reported Self-Confidence (0=very low confidence to 100=very high confidence) before Discharge Testing on Five VAD Skills.
Time Frame: 3 months
Population: patients and caregiver who completed training through hospital discharge
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Traditional VAD Training (Patients) | Traditional VAD Training (Caregivers) | Simulation-based VAD Training (Patients) | Simulation-based VAD Training (Caregivers)
Number analyzed (Participants) | 25 | 25 | 24 | 24
score on a scale
  VAD Driveline exit site sterile dressing changes | 40 [10 to 65] | 90 [75 to 100] | 50 [0 to 87.5] | 100 [90 to 100]
  Changing the VAD controller during emergencies | 90 [72.5 to 100] | 100 [90 to 100] | 95 [80 to 100] | 100 [92.5 to 100]
  Changing power sources on the VAD | 100 [92.5 to 100] | 100 [95 to 100] | 100 [90 to 100] | 100 [100 to 100]
  Troubleshooting emergency VAD-related malfunction | 90 [80 to 100] | 90 [70 to 100] | 90 [80 to 100] | 95 [72.5 to 100]
  Recognizing VAD-specific signs and symptoms | 100 [80 to 100] | 100 [75 to 100] | 100 [92.5 to 100] | 100 [90 to 100]

ADVERSE EVENTS:
Time Frame: 1 year post patient discharge
Description: NOTE: All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed in "Traditional VAD Training (Caregivers)" and "Simulation-based VAD Training (Caregivers)" participants because they are not followed clinically as part of this study.
Arm/Group | Traditional VAD Training (Patients) | Simulation-based VAD Training (Patients)
All-Cause Mortality (participants affected / at risk) | 10/33 | 10/36
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/36
Other Adverse Events (participants affected / at risk) | 0/33 | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-03): https://cdn.clinicaltrials.gov/large-docs/05/NCT03073005/Prot_SAP_000.pdf